CLINICAL TRIAL: NCT07387874
Title: Trastuzumab Rezetecan Alone or in Combination for the Treatment of Patients With Recurrent or Metastatic Malignant Solid Tumors Expressing HER-2 Protein: A Single-Center, Real-World Study
Brief Title: A Real-World Study of Trastuzumab Rezetecan in HER2+ Solid Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Lixiaoling (Other)
Responsible Party: Sponsor-Investigator, Lixiaoling, Chief Physician, Beidahuang Industry Group General Hospital
Organization: Beidahuang Industry Group General Hospital (Other)
Other Study IDs: SHR-A1811-HLJ-002
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Recurrent or Metastatic Solid Tumors
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment arm: Trastuzumab Rezetecan: ± Other Drugs
  Interventions: Drug: Trastuzumab Rezetecan; Drug: Other Drugs

INTERVENTIONS:
Drug: Trastuzumab Rezetecan — Trastuzumab Rezetecan: 4.8 mg/kg, administered every 21 days as one treatment cycle. Patients will receive treatment according to the investigator-defined regimen containing Trastuzumab Rezetecan until disease progression (PD), intolerable toxicity, patient-initiated withdrawal, or the occurrence of other medical events determined by the physician that make the combination therapy unsuitable for continuation.
Drug: Other Drugs — The administration regimens for Trastuzumab Rezetecan include, but are not limited to:
  Combination with immune checkpoint inhibitors ± other agents Combination with targeted agents ± other agents Combination with radiotherapy ± other agents

SUMMARY:
To Observe and Evaluate the Safety Profile of Trastuzumab Rezetecan Alone or in Combination in Patients with HER-2 Protein-Expressing Recurrent or Metastatic Malignant Solid Tumors in a Real-World Setting.

DETAILED DESCRIPTION:
Trastuzumab Rezetecan specifically binds to HER2 on the surface of tumor cells. The conjugate is subsequently internalized into the cells and transported to lysosomes, where the linker is cleaved by cathepsins to release the free toxin SHR169265. This payload inhibits the activity of DNA topoisomerase I, thereby inducing apoptosis in tumor cells. Owing to the high membrane permeability of SHR169265, a bystander killing effect is also observed: after being released inside tumor cells, it can diffuse into neighboring cells, exerting cytotoxic effects even on HER2-negative cells. This study aims to evaluate the efficacy and safety of Trastuzumab Rezetecan, either as monotherapy or in combination regimens, in patients with HER2-expressing recurrent or metastatic malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and agree to participate in this study.
2. Histologically or cytologically confirmed diagnosis of advanced solid tumor.
3. Age ≥ 18 years.
4. HER2 protein expression (including IHC 1+, IHC 2+, IHC 3+, or IHC 0 with ≤10% of invasive tumor cells showing incomplete/weak membrane staining). HER2 protein expression test results must be within 2 years.
5. Patients with advanced solid tumors who have failed, are intolerant to, or refuse standard therapy, and are deemed by the investigator as suitable to receive Trastuzumab Rezetecan monotherapy or combination therapy.

Exclusion Criteria:

1. Patients who are concurrently receiving other therapies of the same class.
2. Patients currently enrolled in another interventional clinical study.
3. Females with confirmed pregnancy or during lactation.
4. Any other condition that, in the opinion of the investigator, renders the patient unsuitable for participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on investigator assessment, patients with HER-2 protein-expressing recurrent or metastatic malignant solid tumors are eligible to receive trastuzumab, either as monotherapy or in combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Safety （Incidence of Grade ≥3 AEs） | From the first dose on Day 1 through the last dose, for up to 3 years
  Safety （Incidence of Grade ≥3 AEs）

SECONDARY OUTCOMES:
ORR | from the date of the first dose to the date of disease progression evaluated based on RECIST v1.1 criteria, or initiation of other anti-tumor treatment, whichever occurs first, up to 6 months
  Overall Response Rate
PFS | From the first vaccination to the first recorded disease progression or death, the assessment period was up to 36 months.
  Progression Free Survival
OS | from the date of the first dose to the date of death for any reason, up to 3 years
  Overall Survival
iORR | From the first dose until the occurrence of intracranial progression or death (whichever occurs first), assessed up to 6 months.
  Intracranial Objective Response Rate
iPFS | From the date of the first dose to the date of the first documented intracranial progression, assessed for up to 3 years.
  Intracranial Progression-Free Survival

OTHER OUTCOMES:
Correlation between HER2 Expression Levels and Safety and Efficacy | from the first drug administration up to 3 years
  Safety and Efficacy According to HER2 Expression Levels (IHC 1+, IHC 2+, IHC 3+, or IHC 0 with ≤10% of Invasive Tumor Cells Showing Incomplete/Weak Membrane Staining)
Safety（ Incidence of AEs and SAEs） | From the first dose on Day 1 through the last dose, for up to 3 years
  Safety（ Incidence of AEs and SAEs）

CONTACTS AND LOCATIONS:
Locations (1):
- BeidahuangGGH, Harbin, China

IPD SHARING:
Plan to Share IPD: No